CLINICAL TRIAL: NCT05271240
Title: A Phase III Randomized Trial of Repeated Superselective Intraarterial Cerebral Infusion (SIACI) of Bevacizumab (Avastin) With Temozolomide and Radiation Compared to Temozolomide and Radiation Alone in Newly Diagnosed Glioblastoma (GBM)
Brief Title: Repeated Superselective Intraarterial Cerebral Infusion (SIACI) of Bevacizumab With Temozolomide and Radiation Compared to Temozolomide and Radiation Alone in Newly Diagnosed GBM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0014
Record Dates: First submitted 2022-02-22; First posted 2022-03-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioma, Malignant; GBM; Brain Cancer; Glioblastoma, IDH-wildtype; Glioblastoma Multiforme, Adult
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — Bevacizumab; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SIACI of Bevacizumab (Avastin) with Temozolomide and Radiation (Experimental): Repeated Superselective Intraarterial Cerebral infusion (SIACI) of Bevacizumab (Avastin) with Temozolomide and Radiation
  Interventions: Drug: Repeated Superselective Intraarterial Cerebral infusion (SIACI) of Bevacizumab (Avastin) with Temozolomide and Radiation
- Standard of care Temozolomide and Radiation (Active Comparator): Standard of care Temozolomide and Radiation
  Interventions: Drug: Temozolomide and Radiation Alone

INTERVENTIONS:
Drug: Repeated Superselective Intraarterial Cerebral infusion (SIACI) of Bevacizumab (Avastin) with Temozolomide and Radiation — Subjects who are assigned to the IA BV+TMZ/RT group (Treatment Group), in addition to your standard of care cancer treatment, you will have a dose of bevacizumab delivered directly to your brain through superselective intra-cranial intra-arterial catheterization of the arteries that supply blood to your brain tumor along with the start of the initial 42 day oral temozolomide treatment. IA BV will be repeated every three months for a total of 3 infusions.
  Other Names: IA BV+TMZ/RT; Intraarterial Bevacizumab
  Arms: SIACI of Bevacizumab (Avastin) with Temozolomide and Radiation
Drug: Temozolomide and Radiation Alone — Subjects who are assigned to the TMZ/RT alone group (Control Group) you will receive standard of care cancer treatment that involves a daily oral dose of temozolomide for 42 days with radiation to the tumor followed by 28 days of rest and then repeated maintenance treatment cycles of daily oral temozolomide 5 days on and 23 days off.
  Other Names: TMZ/RT alone
  Arms: Standard of care Temozolomide and Radiation

SUMMARY:
Primary brain cancer kills up to 10,000 Americans a year. These brain tumors are typically treated by surgery, radiation therapy and chemotherapy, either individually or in combination. Present therapies are inadequate, as evidenced by the low 5-year survival rate for brain cancer patients, with median survival at approximately 12 months. Glioma is the most common form of primary brain cancer, afflicting approximately 7,000 patients in the United States each year. These highly malignant cancers remain a significant unmet clinical need in oncology.

The investigators have completed a Phase I clinical trial that has shown that Superselective Intraarterial Cerebral Infusion (SIACI) of Bevacizumab (BV) is safe up to a dose of 15mg/kg in patients with recurrent malignant glioma. Additionally, the investigators have shown in a recently completed Phase I/II clinical trial, that SIACI BV improves the median progression free survival (PFS) from 4-6 months to 11.5 months and overall survival (OS) from 12-15 months to 23 months in patients with newly diagnosed GBM. Therefore, this two-arm, randomized trial (2:1) is a follow up study to these trials and will ask simple questions: Will this repeated SIACI treatment regimen increase progression free survival (PFS-primary endpoint) and overall survival (OS-secondary endpoint) when compared with standard of care in patients with newly diagnosed GBM? Exploratory endpoints will include adverse events and safety analysis as well as quality of life (QOL) assessments. The investigators expect that this project will provide important information regarding the utility of repeated SIACI BV therapy for newly diagnosed GBM and may alter the way these drugs are delivered to our patients in the near future.

DETAILED DESCRIPTION:
Those randomized to the treatment group (IA BV+TMZ/RT )the experimental aspects will include:

1. Subjects will first be treated with Mannitol prior to IA BV infusion. Mannitol is delivered IA, 12.5 mL over 2 minutes in order to disrupt the blood brain barrier. IA mannitol has been used in several thousand patients in previous studies for the IA delivery of chemotherapy for malignant glioma.
2. Subjects will then be treated with repeated IA BV. Each patient will receive one dose of IA BV on day 30, followed by chemoradiation. IA BV will be repeated every three months for a total of 3 infusions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female 18 years of age or older.
2. Subject has a confirmed diagnosis of GBM according to the 2021 WHO Classification of Tumors of the CNS. Accordingly, eligible GBM patients will comprise only IDH-wild type astrocytomas with microvascular proliferation or necrosis or one or more of 3 genetic parameters (TERT promoter mutations, EGFR gene amplification, or combined gain of entire chromosome 7 and loss of entire chromosome 10).
3. Subject has a Karnofsky Performance Status (KPS) 70% or greater.
4. Subject has a life expectancy of at least 6 months, in the opinion of the Investigator.
5. Subject must be able to undergo MRI evaluation.
6. Subject meets the following laboratory criteria:

   i. White blood count ≥ 3,000/μL ii. Absolute neutrophil count ≥ 1,500/μL iii. Platelets ≥ 100,000/μL iv. Hemoglobin > 10.0 g/dL (transfusion and/or ESA allowed) v. Total bilirubin and alkaline phosphatase ≤ 2x institutional upper limit of normal (ULN) vi. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN vii. Blood urea nitrogen (BUN) and creatinine < 1.5 x ULN
7. Females of reproductive potential must have a negative serum pregnancy test and be willing to use an acceptable method of birth control.
8. Males of reproductive potential must be willing to use an acceptable method of birth control to ensure effective contraception with partner.
9. Able to understand and willing to sign an institutional review board (IRB)-approved written informed consent document (legally authorized representative permitted).

Exclusion Criteria:

1. Subject has initiated chemotherapy or radiation treatment for diagnosis of or GBM.
2. Subject has an IDH mutant astrocytoma or other non GBM brain tumor according to the 2021 WHO classification of Tumors of the CNS.
3. Subject intends to participate in another clinical trial
4. Subject has an active infection requiring treatment.
5. Subject has radiographic evidence of multi-focal disease or leptomeningeal dissemination.
6. Subject has a history of other malignancy unless the patient has been disease-free for at least 5 years. Adequately treated basal cell carcinoma or squamous cell skin cancer is acceptable regardless of time, as well as localized prostate carcinoma or cervical carcinoma in situ after curative treatment
7. Subject has a known positive test for human immunodeficiency virus infection, or active hepatitis B or hepatitis C infection.
8. Subject has a history or evidence of any other clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
9. Subject, if female, is pregnant or is breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 62 months
  The primary end point will be overall survival (OS). Overall survival is defined as the time from randomization until death due to any cause. Participants who are still alive at the time of analysis will be censored at their last known alive date.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 62 months
  The secondary end point will be progression-free survival (PFS). PFS is defined from the time of randomization until first documentation of disease progression (according to RANO Criteria), or death from any cause, whichever occurs first. Participants without documented disease progression at the time of analysis will be censored at the time of their last tumor assessment.

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Feinstein Institute for Medical Research/Lenox Hill Hospital
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States